CLINICAL TRIAL: NCT03536897
Title: Intraoperative Radiation Therapy (IORT) Following Breast Conserving Surgery for Early Stage Breast Cancer Registry
Brief Title: IORT Following Breast Conserving Surgery for Early Stage Breast Cancer Registry
Status: Recruiting | Type: Observational
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 180212-1
Record Dates: First submitted 2018-05-07; First posted 2018-05-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; invasive ductal carcinoma; intraoperative radiation therapy; iort
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- IORT: All patients will undergo a partial mastectomy with sentinel lymph node biopsy with the goal of achieving a margin-negative resection while maintaining good cosmetic outcome. Immediately following partial mastectomy and frozen section evaluation of the sentinel lymph nodes, IORT is to be delivered. Intraoperative radiation therapy will involve 50 kV xrays to a dose of 20 Gy during breast conserving surgery. After surgery, patients are followed based on the standard schedule determined by their surgeon for 5 years.
  Interventions: Radiation: IORT

INTERVENTIONS:
Radiation: IORT — Intraoperative radiation therapy with INTRABEAM system to a dose of 20 Gy

SUMMARY:
This is a prospective, registry trial which will enroll women aged 65 and above with early stage, low risk breast cancer who will be treated with partial mastectomy and intraoperative radiation therapy (IORT). The primary aim is to determine the 5-year risk of in-breast tumor recurrence. Secondary aims include identification of acute- and late-toxicity, cosmetic result, disease-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ECOG performance status 0-1
* Age 65 years or older
* cT1 or cT2 (≤3.0 cm)
* Invasive ductal carcinoma histology
* Estrogen receptor positive (ER+)
* Grade 1 or Grade 2
* Clinically negative lymph nodes (cN0) by examination, imaging and/or nodal sampling
* Suitable for breast conserving surgery and radiation therapy
* Patient must be able to provide study-specific informed consent

Exclusion Criteria:

* Multi-centric cancer not amenable to single lumpectomy
* Prior ipsilateral whole breast radiation
* Known BRCA 1 or BRCA 2 mutation
* Status post neoadjuvant hormonal or chemotherapy
* Invasive lobular histology
* Pure ductal carcinoma in situ (DCIS)
* Grade 3
* Diffuse suspicious microcalcifications

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Women aged 65 and above with early stage breast cancer, ER+, low to intermediate grade invasive ductal carcinoma of the breast amenable to breast conserving surgery and radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2028-02-27 (Estimated); Study Completion 2028-02-27 (Estimated)

PRIMARY OUTCOMES:
In-Breast Tumor Recurrence (IBTR) | 5 years
  Ipsilateral In-Breast Tumor Recurrence (IBTR): defined as biopsy-proved invasive or in situ breast cancer (except LCIS) in the ipsilateral breast.

SECONDARY OUTCOMES:
Late Toxicity | 5 years
  Degree of late radiation toxicity will be scored based upon RTOG/EORTC (Radiation Therapy Oncology Group/Eastern Oncology Radiation Therapy Consortium) late radiation morbidity scoring schema for subcutaneous tissue as well as cosmetic result.
  The RTOG/EORTC late radiation morbidity scoring schema on subcutaneous tissue is as follows:
  * GRADE 1: Slight induration (fibrosis) and loss of subcutaneous fat
  * GRADE 2: Moderate fibrosis but asymptomatic; slight field contracture; <10% linear reduction
  * GRADE 3: Severe induration and loss of subcutaneous tissue; field contracture > 10% linear measurement
  * GRADE 4: Necrosis
Acute Toxicity | 3 months
  Acute radiation toxicity will be scored at the first follow-up visit after IORT (4-6 weeks after treatment).
  Radiation dermatitis will be scored based upon CTCAE (Common Terminology Criteria for Adverse Events) v4.03 scale as follows:
  * GRADE 1: Faint erythema or dry desquamation
  * GRADE 2: Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin folds and creases; moderate edema
  * GRADE 3: Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion
  * GRADE 4: Life threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated
  Other acute toxicity will also be scored per the CTCAE v4.03 scale and will be rated on the relation to radiation therapy (definitely related, probably related, possibly related, unlikely related, unrelated)
Disease Free Survival | 5 yeras
  Disease Free Survival
Overall Survival | 5 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Malolan Rajagopalan, MD, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel West Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No